CLINICAL TRIAL: NCT03763058
Title: The Effect of Music Therapy on Episodic Migraine Patients Under the Care of Chronic Pain Department - A Pilot Trial
Brief Title: Music Intervention on Migraine Headaches
Acronym: CHU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association de Musicothérapie Applications et Recherches Cliniques (Other)
Collaborators: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MusicMig
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Results first posted 2019-07-18 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Migraine Headache
Keywords: Migraine; Headache; Music intervention; Pain; Smartphone application
MeSH Terms: conditions — Migraine Disorders; Headache; Pain | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: A monocentric prospective before-after study on patients carried out in chronic pain department of the CHU Sud Reunion. Patients will be evaluated for inclusion in the study, and will complete the 3-month music intervention. Participants will complete 1-2 sessions of listening to music per day, with a minimum of 15 sessions per month. Before starting the musicotherapy program, retrospective data will be collected on the month prior regarding migraine attacks (frequency, severity, duration, treatment intake).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music intervention (Other): The music intervention is administered via a smartphone- (and computer-) based application called Music Care.
  Interventions: Other: Music Therapy

INTERVENTIONS:
Other: Music Therapy — The music intervention is administered via a smartphone- (and computer-) based application called Music Care. The Music Care app is a receptive music intervention, allowing the patient to freely adjust the length of and choose the preferred style between different sequences of instrumental music. All musical pieces were recorded in high-quality recording studios with professional musicians. Music Care utilizes the "U" technique designed to gradually relax the listener. The "U" technique is implemented using a musical sequence of 20 minutes that was divided into 5 different musical pieces at 3 to 4 minutes each.
  Participants will complete 1-2 sessions of listening to music per day, with a minimum of 15 sessions per month.

SUMMARY:
Migraine is a frequent pathology, highly linked to anxio-depressive factors. Non-drug approaches are part of the therapeutic arsenal. Music therapy is a recent discipline expanding in hospital services and specialised ambulatory centers. The main objective of this study is to assess the effect of " U " technique in receptive music therapy on migraine frequency, on patients suffering from episodic migraines, through " Music care " software home use. Secondary objectives are to assess this technique impact on migraine intensity, duration, emotional effect (HAD score), functional impact (HIT-6 score), and acute treatment administration. This is a monocentric prospective before-after study carried out in chronic pain department of the CHU Sud Reunion.

DETAILED DESCRIPTION:
Despite converging evidence that music interventions are beneficial in a number of pain domains, additional research is needed to understand the impact of a music intervention on the debilitating nature of migraine headaches. Interestingly, a recently developed smartphone application called Music Care has been introduced as a music-intervention tool; however music type is controlled by the individual. A patient-controlled music intervention administered by Music Care has shown to alleviate negative psychological (e.g., depression) and physiological (e.g., pain and discomfort) outcomes associated with general chronic pain. However, no study has examined how music interventions administered via Music Care may be beneficial for individuals who experience migraines, thus potentially highlighting the effects of receptive music techniques in music therapy.

Therefore, the present investigation sought to examine the potential benefits of a patient-controlled, 3-month music intervention in individuals diagnosed with migraine headaches using the Music Care application. Patients from the university hospital center Sud Reunion (Saint Pierre, Reunion Island, France) within the Chronic Pain Consultation Group will be evaluated for inclusion in the study and will complete the 3-month music intervention. Participants will complete 1-2 sessions of listening to music per day, with a minimum of 15 sessions per month.

The following measures will be collected: the frequency of migraine attacks, the average duration of migraine attacks and the average intensity of migraine attacks. Patients will also rate levels of anxiety and depression associated with migraine headaches via the Hospital Anxiety and Depression Scale (HAD). The impact migraines have on everyday level of functioning will be evaluated using the Headache Impact Test (HIT-6).

This is a pilot study, non-randomized, single arm and single center study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with episodic migraine with at least 4 attacks per month
* Patients with migraines with or without aura with diagnostic criteria per International Headache Society
* Patients with a migraine for more than one year
* Diagnosis age < 50 years
* Patients with an available internet connexion to access Music Care application
* Patients with minimal knowledge in informatics
* Patients who sign their inform consent

Exclusion Criteria:

* Patients aged less than 18 years
* Patients with chronic migraine
* Patients with epilepsy
* Patients with a deficiency on auditive function
* Patients with a disease that could be fatal within the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guilhem PARLONGUE, PhD, Principal Investigator
Locations (1):
- CHU de la Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No
This is not planned to share individual subjects data to other people.

REFERENCES:
- [Result] Guetin S, Ginies P, Siou DK, Picot MC, Pommie C, Guldner E, Gosp AM, Ostyn K, Coudeyre E, Touchon J. The effects of music intervention in the management of chronic pain: a single-blind, randomized, controlled trial. Clin J Pain. 2012 May;28(4):329-37. doi: 10.1097/AJP.0b013e31822be973. PMID 22001666
- [Result] Guetin S, Portet F, Picot MC, Defez C, Pose C, Blayac JP, Touchon J. [Impact of music therapy on anxiety and depression for patients with Alzheimer's disease and on the burden felt by the main caregiver (feasibility study)]. Encephale. 2009 Feb;35(1):57-65. doi: 10.1016/j.encep.2007.10.009. Epub 2008 Feb 20. French. PMID 19250995
- [Result] Meister M, Einsle R, Brunner J, Rhyner K. [Psychofonia--a neurophysiologic music therapy in migraine]. Praxis (Bern 1994). 1999 May 20;88(21):946-9. German. PMID 10412281
- [Result] Koenig J, Oelkers-Ax R, Kaess M, Parzer P, Lenzen C, Hillecke TK, Resch F. Specific music therapy techniques in the treatment of primary headache disorders in adolescents: a randomized attention-placebo-controlled trial. J Pain. 2013 Oct;14(10):1196-207. doi: 10.1016/j.jpain.2013.05.006. Epub 2013 Jul 19. PMID 23876282
- [Result] Oelkers-Ax R, Leins A, Parzer P, Hillecke T, Bolay HV, Fischer J, Bender S, Hermanns U, Resch F. Butterbur root extract and music therapy in the prevention of childhood migraine: an explorative study. Eur J Pain. 2008 Apr;12(3):301-13. doi: 10.1016/j.ejpain.2007.06.003. Epub 2007 Jul 30. PMID 17659990

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in Groupe Hospitalier Sud Réunion between 3-15 December 2018.
Pre-assignment Details: Thirty-two patients were screened but not enrolled and assigned to music intervention as they did not fill the inclusion/exclusion criteria.
Groups:
- Music Intervention: The music intervention is administered via a smartphone- (and computer-) based application called Music Care.
  Music Therapy: The music intervention was administered via a smartphone- (and computer-) based application called Music Care. The Music Care app is a receptive music intervention, allowing the patient to freely adjust the length of and choose the preferred style between different sequences of instrumental music. All musical pieces were recorded in high-quality recording studios with professional musicians. Music Care utilizes the "U" technique designed to gradually relax the listener. The "U" technique is implemented using a musical sequence of 20 minutes that was divided into 5 different musical pieces at 3 to 4 minutes each.
  Participants completed 1-2 sessions of listening to music per day, with a minimum of 15 sessions per month.
Period: Overall Study
Arm/Group | Music Intervention
Started | 20
Completed | 18
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Music Intervention
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 42 [19 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Réunion | 20

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Migraine Attacks (Number of Days Per Month)
Description: All data related to migraine like frequency, duration, severity are to be collected in a diary questionnaire. Per ANAES (Agence nationale de l'accréditation et de l'évaluation en santé) recommendations, this means reduction of 50% on frequency of migraine attacks after 3-month treatment period. Comparison will be done between the number of days in the month prior the first music intervention and the number of days in the 3rd month of intervention.
Time Frame: 1 month prior to intervention (pre-treatment) up to 3 months (post-treatment)
Measure: Mean (Standard Deviation); unit: Number of migraine per months
Arm/Group | Music Intervention
Number analyzed (Participants) | 20
Number of migraine per months
  Pre-treatment | 8.45 (3.03)
  Post-treatment | 5.65 (3.73)
Statistical Analysis 1: Comparison: Music Intervention; Test type: Superiority; p = 0.012, Sign test; Mean Difference (Final Values) = -2.8, Standard Deviation 4.19

2. Secondary Outcome: Duration of Migraine Attacks (Hours)
Description: The outcome is the mean duration of migraine attacks per month. Comparison will be done between the month prior the first music intervention and the 3rd month of intervention. The mean duration is calculated by summing the total duration during the month divided by the number of attacks in the month.
Time Frame: 1 month prior to intervention (pre-treatment) up to 3 months (post-treatment)
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Music Intervention
Number analyzed (Participants) | 20
Hours
  Pre-treatment | 10.95 (16.84)
  Post-treatment | 5.5 (7.47)
Statistical Analysis 1: Comparison: Music Intervention; Test type: Superiority; p = 0.002, Sign test; Mean Difference (Final Values) = -5.45, Standard Deviation 15.52

3. Secondary Outcome: Number of Migraine Episodes With Severe Intensity
Description: This data is collected as mild, moderate or severe. The same analysis as the primary outcome will be done by severity. So the frequency of migraine attacks will be compared for each severity.
Time Frame: 1 month prior to intervention (pre-treatment) up to 3 months (post-treatment)
Population: Number of episodes with varying intensity (mild, moderate, severe). Only severe are reported.
Measure: Mean (Standard Deviation); unit: Number of episodes
Arm/Group | Music Intervention
Number analyzed (Participants) | 20
Number of episodes
  Pre-treatment | 2.9 (3.81)
  Post-treatment | 1.7 (1.72)
Statistical Analysis 1: Comparison: Music Intervention; Test type: Superiority; p = 0.045, Sign test; Mean Difference (Final Values) = -1.2, Standard Deviation 2.71

4. Secondary Outcome: Impact of Migraines on Everyday Level of Functioning
Description: This outcome will be evaluated using the Headache Impact Test (HIT-6) score. The total score range is 36-78. A higher score indicates a worse impact of migraines on daily life. Comparison will be done between the score obtained before first music session and at the evaluation done after 3 months of music intervention.
Time Frame: 1 month prior to intervention (pre-treatment) up to 3 months (post-treatment)
Population: Difference between post and pre-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Music Intervention
Number analyzed (Participants) | 20
score on a scale
  Pre-treatment | 62.75 (6.12)
  Posttreatment | 59.1 (6.78)
Statistical Analysis 1: Comparison: Music Intervention; Test type: Superiority; p < 0.001, Sign test; Mean Difference (Final Values) = -3.65, Standard Deviation 4.59

5. Secondary Outcome: Reduction on Anxiety and Depression
Description: This outcome will be evaluated using Hospital Anxiety and Depression Scale (HAD). The total scores range is 0-21 for both depression and anxiety scores. A higher score indicates a worse depression and anxiety. Comparison will be done between the score obtained before first music session and at the evaluation done after 3 months of music intervention.
Time Frame: 1 month prior to intervention (pre-treatment) up to 3 months (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Music Intervention
Number analyzed (Participants) | 20
score on a scale
  Anxiety HAD pre-treatment | 9.05 (3.75)
  Anxiety HAD post-treatment | 7.4 (3.79)
  Depression HAD pre-treatment | 6.45 (3.88)
  Depression HAD post-treatment | 4 (3.46)
Statistical Analysis 1: Comparison: Music Intervention; Total HAD score; Test type: Superiority; p < 0.001, Sign test; Mean Difference (Final Values) = -4.15, Standard Deviation 5.1

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Music Intervention
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
* No control group
* Future studies to explore music intervention compared to other therapeutic options
* results to be interpreted with caution as headache symptoms are self-collected

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT03763058/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT03763058/SAP_001.pdf